CLINICAL TRIAL: NCT01527812
Title: Optimal Positioning of Local Anaesthetic in Femoral Nerve Block Prior to Operative Fixation of Fractured Neck of Femur
Brief Title: Optimal Positioning of Local Anaesthetic in Femoral Nerve Block Prior to Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Szilard Szucs, Clinical Tutor in Anaesthesia, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECM 4 (zz) 08/12/09; ECM 4 (zz) 08/12/09 (Other: Clinical Research Ethics Committee of the Cork Teaching Hospitals)
Record Dates: First submitted 2012-02-01; First posted 2012-02-07 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-02

CONDITIONS: Fractured Neck of Femur
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Above the femoral nerve (Experimental): In Group I we will inject the local anaesthetic below the fascia iliaca and above the femoral nerve.
  Interventions: Procedure: Femoral nerve block
- Below the femoral nerve (Experimental): In Group II we will inject the local anaesthetic below the femoral nerve and above the fascia of the iliopsoas muscle.
  Interventions: Procedure: Femoral nerve block
- Circumferential (Experimental): In Group III a circumferential spread will be achieved with multiple injections.
  Interventions: Procedure: Femoral nerve block

INTERVENTIONS:
Procedure: Femoral nerve block — We will perform an ultrasound guided femoral nerve block. For locating the nerve a 5 cm, 6-13 MHz linear probe (Sonosite Turbo M, Bothwell WA, USA) will be used. After the examination of the anatomy of the femoral artery we will fix the probe transversal to the thigh below the inguinal crease and above the ramification of deep femoral artery and make skin marks on this position. A 22 G 50 mm long Stimuplex BBraun needle will be used. 15 ml 2 % lignocaine will be injected.

SUMMARY:
The aim of the study is to compare patient comfort and analgesic efficacy of ultrasound guided femoral nerve block using the following endpoints: circumferential spread, anterior or posterior local anaesthetic deposition prior to positioning for spinal anaesthesia for operative fixation of fractured neck of femur.

DETAILED DESCRIPTION:
Fractured neck of femur is a common cause of admission to hospital in elderly patients and requires operative fixation. The recommended anaesthetic technique for these cases is spinal anaesthesia, which is performed with the patient in lateral decubitus. Positioning the patient prior to administering spinal anaesthesia is the most painful manouvre due to the movement of the fractured bone.

Regional anaesthesia is effective in alleviating pain due to trauma, and it has the advantage of producing localized but complete pain relief (1). Femoral nerve blockade prior to positioning for spinal anaesthesia provides excellent pain relief and is a well tolerated procedure (2-5).

Using ultrasound guided femoral nerve block is a relative new method to improving the block success rate. It is widely used in our hospital. In a recent study Casati and al. showed a 42 % decrease of ED50% using ultrasound for localization of the femoral nerve (6). In a recent editorial by Brian D. Sites was mentioned that the positioning of the local anaesthetic in ultrasound guided blocks is unclear (7). We currently follow different patterns in relation to injection of the local anaesthetic solution around the femoral nerve. One of them is a circumferencial spread around the nerve. This, however, needs several needle passes which are likely to be painful for the patient. Another option is injecting the local anaesthetic on one side, above or below the nerve without changing the position of the tip of the needle, avoiding patient discomfort. Whether this results in a comparable quality of sensory block is unknown. The femoral nerve is separated in branches at this level and we assume that the spread of local anaesthetic may influence the quality and the distribution of the block. We propose to study the characteristics of femoral nerve block in relation to different patterns of local anaesthetic injection (circumferencial, inferior or superior).

ELIGIBILITY:
Inclusion Criteria:

* Fractured neck of femur surgical fixation performed under spinal anaesthesia
* ASA I to III

Exclusion Criteria:

* Patient refusal
* Coagulation disorders
* Head injury or other associated injuries
* Previous vascular surgery in the femoral area.
* Loss of consciousness and signs of acute coronary syndrome
* Mini-Mental Score < 25 (see appendix 3)
* Allergy to lignocaine,
* Skin lesions/infection at site of injection
* Sepsis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Verbal rating scale (VRS) pain scores after positioning the patient to performing the spinal anaesthesia. | The patient will be assessed in every five minutes up to 30 minutes after the femoral nerve block.
  Independent blinded observer will assess the patient in the first 30 minutes, in every 5 minute. Sensory perception will be assess by using cold spray in the area of the terminal branch of femoral nerve.
  We will assess the pain on passive movement of the limb (elevating 30 degree) using verbal rating scale (VRS) pain score 1-10. When the patient reports less than 4 at the VRS the patient will be positioned for spinal anaesthesia.
  If the threshold isn't achieved by 30 minutes, the block will be classified as failure. Additional opioid medication and/or sedation will be administered.

SECONDARY OUTCOMES:
Sensory distribution of the nerve block. | The patient will be assessed in every five minutes up to 30 minutes after the femoral nerve block.
  An independent blinded observer (not present during block placement) will assess in the first 30 minutes (at 5 minute intervales) the sensory nerve block using a modified Bromage score. Sensory perception will be assessed using cold (ethyl chloride spray) in the area of the vastus medialis, vastus intermedius, vastus lateralis and saphenous nerve innervation area (terminal branch of femoral nerve).
Number of needle passes | during performing the femoral nerve block
  The Anaesthestist who performing the femoral nerve block was asked how many needle passes needed for the femoral nerve block.
Femoral nerve block onset time | In the first 30 minutes after the femoral nerve block
  We will assess the pain on passive movement of the limb (elevating 30 degree from the initial positioning) using verbal rating scale (VRS) pain score 1-10. When the patient reports less than 4 at the VRS the sensory block will be deemed adequate and the patient will be positioned on the side for spinal anaesthesia.
Patient satisfaction | After the surgery in the recovery area before the patient will be discharged to the ward.
  After the surgery during the recovery time, we will ask the patients regarding there Satisfaction, will be used visual analog scale 0-100 mm for measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Szilard Szucs, MD, Principal Investigator — Cork University Hospital, Ireland
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

REFERENCES:
- [Derived] Szucs S, Morau D, Sultan SF, Iohom G, Shorten G. A comparison of three techniques (local anesthetic deposited circumferential to vs. above vs. below the nerve) for ultrasound guided femoral nerve block. BMC Anesthesiol. 2014 Jan 25;14:6. doi: 10.1186/1471-2253-14-6. PMID 24460975